CLINICAL TRIAL: NCT00302939
Title: Studies in the Etiology of Anemia in an Unselected Sequential Referral Population
Brief Title: Etiology of Anemia
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: William B. Ershler, M.D., Principle Investigator, National Institute on Aging
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0062
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2010-04

CONDITIONS: Anemia
Keywords: Aging
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow aspirate, urine, blood serum

SUMMARY:
This study looks at the causes of anemia in adults of all ages who are referred by their primary care physician.

DETAILED DESCRIPTION:
This study is being done to determine if the range of causes of anemia changes with advancing age. The goal of this study is to apply research methods to see if causes of anemia can be determined in patients where a clear cause is not found with routine clinical testing available to all patients in physician offices.

Participants in this study will be evaluated at the NIA-ASTRA unit at Harbor Hospital in Baltimore. Testing will consist of both diagnostic and research blood and urine testing along with history and physical exam. An optional bone marrow aspirate or aspirate and biopsy may be performed if the patient permits and it is indicated for either research or clinical diagnostic purposes. All study information supporting a specific diagnosis will be provided to the patient and, at their request, to their primary care physician if specific treatment is indicated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Hemoglobin (Hgb) less than 13 in males and females

Exclusion Criteria:

* Pregnant or nursing women
* Participation within the past six weeks in another research study which the Principal Investigator believes is incompatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Ershler, MD, Principal Investigator — NIA/NIH
Locations (1):
- National Institute on Aging, Baltimore, Maryland, United States

REFERENCES:
- [Background] Guralnik JM, Eisenstaedt RS, Ferrucci L, Klein HG, Woodman RC. Prevalence of anemia in persons 65 years and older in the United States: evidence for a high rate of unexplained anemia. Blood. 2004 Oct 15;104(8):2263-8. doi: 10.1182/blood-2004-05-1812. Epub 2004 Jul 6. PMID 15238427
- [Background] Artz AS, Fergusson D, Drinka PJ, Gerald M, Bidenbender R, Lechich A, Silverstone F, McCamish MA, Dai J, Keller E, Ershler WB. Mechanisms of unexplained anemia in the nursing home. J Am Geriatr Soc. 2004 Mar;52(3):423-7. doi: 10.1111/j.1532-5415.2004.52116.x. PMID 14962159